CLINICAL TRIAL: NCT02279680
Title: The Associative Memory in Autism Spectrum Disorders Without Intellectual Disability
Brief Title: Associative Memory in Adults With an Autism Spectrum Disorder
Acronym: MEM-T2A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-AO1800-45
Record Dates: First submitted 2014-06-23; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Other): Adults between 18 and 30 years old right handing Patients with ASD
  Interventions: Device: Electroencephalography; Behavioral: Neuropsychological assesments
- Healthy volunteers (Other): Adults between 18 and 30 years old Right handing Healthy
  Interventions: Device: Electroencephalography; Behavioral: Neuropsychological assesments

INTERVENTIONS:
Device: Electroencephalography
Behavioral: Neuropsychological assesments

SUMMARY:
The objective of this multidisciplinary project is to explore the deficit of associative memory in ASD (Autistic Spectrum Disorder) that could result from abnormal brain connectivity. The hypothesis of abnormal functioning of the fronto-hippocampal network has been evocated but has never been tested. Hence, the present project will include two complementary assessments conducted on a group of adults aged from 18 to 30 with ASD compared to a control group matched in chronological age and intellectual quotient. The first assessment is devoted to the study of associative memory and its EEG correlates and the second focused on the investigation of perceptual strategies related to associative memory using the technique of Eye-tracking. Both behavioral and imaging data would provide new insights on the relationship between perception and memory in ASD.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 30 years old
* right handed
* affiliated to the french national health care system
* ASD only for the group of patients

Exclusion criteria :

* mental retardation
* schizophrenia
* ADHD
* brain injury with lost of consciousness
* neurological disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The associative memory index | 2 years

SECONDARY OUTCOMES:
theta and gamma oscillations during the associative memory task | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc BALEYTE, PU-PH, Principal Investigator — University Hospital, Caen
Locations (1):
- UMR1077 Inserm/EPHE/UCBN, Caen, Caen, France